CLINICAL TRIAL: NCT02636634
Title: Non Invasive Methods for Differential Diagnosis Radionecrosis/Recurrence After Radiosurgery of Brain Metastases. CV-METANEC
Brief Title: Non Invasive Methods for Differential Diagnosis Radionecrosis/Recurrence After Radiosurgery of Brain Metastases
Acronym: CV-METANEC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P071243; 2009-014458-14 (EudraCT Number)
Record Dates: First submitted 2015-12-08; First posted 2015-12-22 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Brain Metastases; Growing Lesions After Radiosurgical Treatment
Keywords: diagnostic strategy; brain metastases; radiation necrosis; relapse; PET-FET and MSR; radiosurgery
MeSH Terms: conditions — Brain Neoplasms; Recurrence | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- diagnostic imaging strategy (Other): PET-FET (positron emission tomography using 1-Fluoro-Ethyl-Tyrosine) and MSR (magnetic resonance spectroscopy) before biopsy
  Interventions: Other: imaging

INTERVENTIONS:
Other: imaging

SUMMARY:
The purpose of this multicenter study is to assess a diagnostic strategy concerning differential diagnosis between radiation necrosis and relapse in brain metastases treated with radiosurgery. Two non-invasive tests - positron emission tomography (PET) with 1F-fluoro-ethyl-tyrosine (FET) and magnetic resonance spectroscopy (MRS) - will be compared to histology in a cohort of patients presenting growing lesions 6 months after radiosurgical treatment.

The results of this study should help to earlier diagnosis of recurrences after radiosurgery and to perform an appropriate treatment for patients.

DETAILED DESCRIPTION:
The purpose of the study is to assess a diagnostic strategy by monitoring brain metastases after radio surgical treatment . Data from two non-invasive techniques: PET-FET (positron emission tomography using 1-Fluoro-Ethyl-Tyrosine) and MSR (magnetic resonance spectroscopy) will be compared to histological examination (gold standard) in patients with active persistent and increased lesion 4 months after radiosurgery. The study should develop a decision-making algorithm based on non-invasive tests and allow improving the length and quality of life of these patients.

Early differential diagnosis between relapse and radio necrosis after radiosurgery would allow:

* To perform resection of tumor relapse
* To treat feasable/inoperable tumor relapse with a salvage radiosurgery
* To avoid irradiation for patients presenting radiation necrosis
* To reduce the corticosteroid prescription period. Validation of non-invasive diagnostic tools should in fine avoid biopsy. In addition, the results of this study should help to better estimate the true incidence of radiation necrosis and better specify the predictors of this complication.

CV-METANEC is a prospective, multicenter, open, multidisciplinary study involving the following departments: neurosurgery, neuroradiology, nuclear medicine and neuropathology.

4 centers participating in the study: Groupe Hospitalier Pitié-Salpêtrière University Hospital, Lariboisière Hospital, Lille University Hospital of Clermont Ferrand and Toulouse University Hospital.

Patients are included if they were treated by radiosurgery for one or more brain metastases. The interval between the radiosurgical treatment and the inclusion is at least 6 months. The lesion is clinically and / or MRI evolving.

The criterion used to measure the discriminating power of the algorithm to rank the differential between recurrences with or without radionecrosis or only radionecrosis is the area under the ROC (receiver operating characteristic) curve. The inclusion of 90 subjects will achieve a standard deviation of the area under the curve 0.04.

The duration of study participation will be five weeks, from inclusion until the end of hospitalization. Subsequently, the patient will be followed as usual.

Inclusion D0: whether the conditions of inclusion are applied, the patient signs the consent form and exams before surgery are planned: SRI-MRI, examination of scintigraphy and anesthesia consultation.

D15: MRI (neuroradiology) and anesthetic consultation (neurosurgery).

D30-D33 (+/- 7 days): 3 days of hospitalization:

D30: MRI / MRS always done before-FET PET D31: stereotactic biopsy for histological samples. D33: CT scan before the patient is discharged. Total study duration: 5 years

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years.
* Patient treated with radiosurgery for one or more brain metastases Free -Intervally between radiosurgical treatment and inclusion in the study at least four months.
* Lesion (S) treated (s) and followed (s) with the criteria for a clinically active lesion (progressive deficit, seizures, intracranial hypertension steroid-dependent) and / or MRI (increased volume of contrast enhancement with peri-lesional edema and mass effect on two successive examinations at 1 month interval).
* Karnofsky index> 50.
* Prognostic compatible for survival with a follow-up at least three months from the date of inclusion.
* Effective contraception for women of childbearing potential or negative pregnancy test within 72 hours.
* Signed informed consent obtain
* Affiliation to the social security system

Exclusion Criteria:

* Contraindication to MRI examination
* Clearance of the creatinine incompatible with the injection of gadolinium
* No potential follow-up in middle or long term
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-06; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
the choline /N-acetyl aspartate ratio at MR spectroscopy | Day 30
the lipid / lactate ratio at MR spectroscopy | Day 30
peak creatine at MR spectroscopy | Day 30
lesional tissue / normal tissue ratio at PET with FET | Day 30
Histological result at biopsy | Day 31
  histology as the gold standard for the diagnostic between radiation necrosis and relapse

CONTACTS AND LOCATIONS:
Overall Officials: Charles-Ambroise VALERY, MD, PhD, Principal Investigator — CHU Pitié-Salpêtrière - Service de Neurochirurgie du Pr Philippe Cornu - Babinsky
Locations (1):
- CHU Pitié-Salpêtrière - Service de Neurochirurgie du Pr Philippe Cornu - Babinsky, Paris, France